CLINICAL TRIAL: NCT02458365
Title: A Stage-Based Expert System for Teen Dating Violence Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44MH086129 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2015-07

CONDITIONS: Violence; Bullying
Keywords: Violence; Bullying; Social skills; Prevention & control; Adolescent
MeSH Terms: conditions — Bullying; Social Skills | interventions — Health; Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teen Choices (Experimental): Teen Choices: A Program for Healthy Nonviolent Relationships
  Interventions: Behavioral: Teen Choices: A Program for Healthy Nonviolent Relationships
- Comparison (Other): Health In Motion
  Interventions: Behavioral: Health In Motion

INTERVENTIONS:
Behavioral: Teen Choices: A Program for Healthy Nonviolent Relationships — A 3-session online, multimedia TTM-based intervention for teen dating violence prevention. For most students, the intervention seeks to reduce risk for dating violence by facilitating progress through the stages of change for using healthy relationship skills; daters are encouraged to use those skills in their dating relationships, and non-daters in their peer relationships, as relationships with peers serve as the foundation for experiences in romantic relationships. For victims of dating violence experiencing fear, the intervention does not focus on healthy relationship skills; instead, it seeks to facilitate progress through the stages of change for keeping oneself safe in relationships.
  Arms: Teen Choices
Behavioral: Health In Motion — A 3-session online, multimedia, TTM-based intervention which targets physical activity, screen time, and healthy eating for obesity prevention. Health In Motion sessions were administered following the baseline, 6-month, and 12-month assessments to increase the benefits of study participation for Comparison schools and students.
  Arms: Comparison

SUMMARY:
Male-to-female intimate partner violence accounts for 26% of violence-related injuries in women presenting in hospital emergency departments and 33% of all female homicides. Adolescence provides an excellent "window of opportunity" for the prevention of intimate partner violence. Patterns of relating in intimate relationships are still relatively undifferentiated and open to influence. However, the evidence supporting traditional, school-based programs for the prevention of teen dating violence is mixed. A major problem with existing programs is that they are "one size fits all," making it difficult to meet the diverse needs of students-boys and girls, individuals who are dating and those who are not, individuals who have experienced dating violence as a victim, perpetrator, or both, and those who have not. Perhaps most importantly, these interventions neglect individual differences in readiness to use healthy, non-violent ways of relating to stay violence-free. In Phase I the objective was to use expert system technology to integrate best practices for teen dating violence prevention with the Transtheoretical Model of Behavior Change (TTM), the "stage model," to develop an interactive, multimedia computer-administered change program that delivers individualized intervention sessions and exercises tailored to stage of change and other individual characteristics. In Phase II, the objective was to complete development of the intervention package and assess its efficacy in a randomized clinical trial involving 3,901 teens from 20 Rhode Island high schools randomly assigned to intervention or comparison. Among youth exposed to risk for dating violence, efficacy was assessed by comparing the intervention and comparison groups on dating violence perpetration and victimization at follow-up. Among youth not exposed to risk for dating violence, efficacy was assessed by comparing intervention and comparison on peer violence perpetration and victimization.

DETAILED DESCRIPTION:
Twenty Rhode Island high schools agreed to participate in the study. A Multiattribute Utility Measurement Approach (Graham, Flay, Johnson, Hansen, & Collins, 1984) was used to ensure that schools assigned to the intervention and comparison conditions were approximately equivalent on school size, student ethnicity, socioeconomic status (SES, percent receiving free or reduced-price lunch), attendance, mobility, truancy, dropout, and standardized test performance. The most similar schools were paired, and one school within each pair was randomly assigned to intervention, and the other to comparison.

The intervention trial was launched in the Fall of 2009. Both the intervention and comparison groups completed a computerized baseline assessment and two follow-up assessments approximately 6 and 12 months later-in the Spring and Fall of 2010. Students assigned to the intervention condition completed their first Teen Choices intervention session immediately following their baseline assessment. The second and third intervention sessions were administered at approximately 1 and 2 months follow-up. Students assigned to the comparison condition completed an alternative evidence-based online TTM-based intervention, Health In Motion, which targets physical activity, screen time, and healthy eating for obesity prevention (Mauriello et al., 2010). Health In Motion sessions were administered following the baseline, 6-month, and 12-month assessments to increase the benefits of study participation for comparison schools and students. Online assessment and intervention sessions were overseen by project research assistants with the assistance of school personnel.

Dating violence outcomes at one year follow-up were were examined in intervention and comparison participants who completed the final assessment and were exposed to risk for dating violence-that is, students who had experienced or perpetrated emotional or physical dating violence in the year prior to the study, who were current daters at baseline, or who dated during the follow-up period. Peer violence outcomes were examined in participants who completed the final assessment and were not exposed to risk for dating violence.

ELIGIBILITY:
Inclusion Criteria:

* Attending one of 20 participating schools
* In grade 9, 10, or 11

Exclusion Criteria:

* Parent submitted opt-out form

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3901 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Levesque, Ph.D., Principal Investigator — Pro-Change Behavior Systems, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Teen Choices: A 3-session online, multimedia TTM-based intervention for teen dating violence prevention. For most students, the intervention seeks to reduce risk for dating violence by facilitating progress through the stages of change for using healthy relationship skills; daters are encouraged to use those skills in their dating relationships, and non-daters in their peer relationships, as relationships with peers serve as the foundation for experiences in romantic relationships. For victims of dating violence experiencing fear, the intervention does not focus on healthy relationship skills; instead, it seeks to facilitate progress through the stages of change for keeping oneself safe in relationships.
- Comparison: Health In Motion: A 3-session online, multimedia, TTM-based intervention which targets physical activity, screen time, and healthy eating for obesity prevention. Health In Motion sessions were administered following the baseline, 6-month, and 12-month assessments to increase the benefits of study participation for Comparison schools and students.
Period: Overall Study
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Started | 2000 | 1901
Completed | 1723 | 1607
Not Completed | 277 | 294

BASELINE CHARACTERISTICS:
Groups:
- Intevention: Teen Choices: A 3-session online, multimedia TTM-based intervention for teen dating violence prevention. For most students, the intervention seeks to reduce risk for dating violence by facilitating progress through the stages of change for using healthy relationship skills; daters are encouraged to use those skills in their dating relationships, and non-daters in their peer relationships, as relationships with peers serve as the foundation for experiences in romantic relationships. For victims of dating violence experiencing fear, the intervention does not focus on healthy relationship skills; instead, it seeks to facilitate progress through the stages of change for keeping oneself safe in relationships.
- Total: Total of all reporting groups
Arm/Group | Intevention: Teen Choices | Comparison: Health In Motion | Total
Number analyzed (Participants) | 2000 | 1901 | 3901
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1989 | 1893 | 3882
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1028 | 988 | 2016
  Male | 972 | 913 | 1885
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 218 | 186 | 404
  Not Hispanic or Latino | 1782 | 1715 | 3497
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 9 | 23
  Asian | 39 | 61 | 100
  Native Hawaiian or Other Pacific Islander | 7 | 12 | 19
  Black or African American | 54 | 107 | 161
  White | 1613 | 1447 | 3060
  More than one race | 72 | 87 | 159
  Unknown or Not Reported | 201 | 178 | 379
Region of Enrollment [Number; unit: participants]
  United States | 2000 | 1901 | 3901

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Perpetrating Physical Dating Violence During Follow-up
Description: A 30-item measure assessing five types of dating violence perpetration and victimization was developed to meet specific needs of this research (Levesque, 2007). Alphas for the five 3-item perpetrator scales are: .88 for emotional mistreatment, .87 for controlling behavior, .91 for threats, .92 for physical violence, and .94 for sexual coercion. At follow-up, in the spring and fall of 2010, the measure assessed dating violence perpetrated and experienced since January 1, 2010. Given the hierarchical structure of the perpetration measure, the emotional mistreatment and controlling behavior scales were combined to represent emotional dating violence perpetration, and the threats, physical violence, and sexual coercion scales were combined to represent physical perpetration. Given extreme non-normal distributions, the two measures were then dichotomized. One or more incidents of physical perpetration during the period in question were coded as "yes," and no incidents as "no".
Time Frame: One year
Population: Participants who were exposed to at least minimal risk for dating violence -- i.e., who had experienced or perpetrated emotional or physical dating violence in the year prior to the study, who were current daters at baseline, or who dated during the follow-up period.
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health in Motion
Number analyzed (Participants) | 1389 | 1216
participants | 240 | 307
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health in Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .62, 95% CI 2-sided [.51 to .75]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health in Motion; Test type: Superiority or Other; p < .0001, Regression, Linear; Adjusted model that controls for potential confounds and covariates, including variables that predicted non-response and the primary outcomes; Odds Ratio (OR) = .55, 95% CI 2-sided [.45 to .68]

2. Secondary Outcome: Number of Participants Experiencing Physical Dating Violence During Follow-up
Description: See above. Cronbach's Alphas for the five victimization scales were .87 for emotional mistreatment, .86 for controlling behavior, .83 for threats, .76 for physical violence, and .90 for sexual coercion. One or more incidents of physical dating violence victimization during the period in question were coded as "yes," and no incidents coded as "no").
Time Frame: One year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 1389 | 1216
participants | 427 | 471
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .70, 95% CI 2-sided [.57 to .84]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .61, 95% CI 2-sided [.50 to .75]

3. Secondary Outcome: Number of Participants Perpetrating Emotional Dating Violence During Follow-up
Description: See above.One or more incidents of emotional dating violence perpetration during the period in question were coded as "yes," and no incidents coded as "no").
Time Frame: One year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 1389 | 1216
participants | 617 | 727
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .53, 95% CI 2-sided [.43 to .67]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .45, 95% CI 2-sided [.36 to .56]

4. Secondary Outcome: Number of Participants Experiencing Emotional Dating Violence During Follow-up
Description: See above.One or more incidents of emotional dating violence victimization during the period in question were coded as "yes," and no incidents coded as "no").
Time Frame: One year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 1389 | 1216
participants | 824 | 903
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .50, 95% CI 2-sided [.41 to .62]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .44, 95% CI 2-sided [.35 to .54]

5. Other Pre Specified Outcome: Number of Participants Perpetrating Physical Peer Violence During Follow-up
Description: Among participants not exposed to risk for dating violence, an 18-item measure assessed three types of peer violence perpetration and victimization (Levesque, 2007). Alphas for the three 3-item perpetrator scales are: .89 for emotional mistreatment, .89 for physical violence, and .94 for sexual coercion. At follow-up, in the spring and fall of 2010, the measure assessed peer violence experienced and perpetrated since January 1, 2010. Given the hierarchical structure of the perpetration measure, the physical violence and sexual coercion scales were combined to represent physical perpetration. One or more incidents of physical perpetration during the period in question were coded as "yes," and no incidents coded as "no".
Time Frame: One year
Population: Participants who were not exposed to at least minimal risk for dating violence (see definition of minimal risk above); among 725 participants not exposed to risk, 44 were inadvertently administered the wrong measures and thus were excluded from analyses, leaving N = 681.
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 324 | 357
participants | 60 | 105
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p = .001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .55, 95% CI 2-sided [.38 to .78]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p = .013, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .60, 95% CI 2-sided [.40 to .90]

6. Other Pre Specified Outcome: Number of Participants Experiencing Physical Peer Violence During Follow-up
Description: See above. Cronbach's Alphas for the three victimization scales were .89 for emotional mistreatment, .89 for physical violence, and .93 for sexual coercion. One or more incidents of physical peer violence victimization during the period in question were coded as "yes," and no incidents coded as "no").
Time Frame: One year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 324 | 357
participants | 105 | 169
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .53, 95% CI 2-sided [.37 to .76]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p = .004, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .54, 95% CI 2-sided [.35 to .82]

7. Other Pre Specified Outcome: Number of Participants Perpetrating Emotional Peer Violence During Follow-up
Description: See above. One or more incidents of peer emotional mistreatment perpetrated during the period in question were coded as "yes," and no incidents coded as "no").
Time Frame: One year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 324 | 357
participants | 157 | 226
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p = .002, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .53, 95% CI 2-sided [.35 to .78]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p = .005, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .50, 95% CI 2-sided [.31 to .81]

8. Other Pre Specified Outcome: Number of Participants Experiencing Emotional Peer Violence During Follow-up
Description: See above. One or more incidents of peer emotional mistreatment experienced during the period in question were coded as "yes," and no incidents coded as "no").
Time Frame: One year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Number analyzed (Participants) | 324 | 357
participants | 198 | 280
Statistical Analysis 1: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p < .0001, Regression, Logistic; Hierarchical logistic regression using random intercepts for school to account for the clustered study design; Odds Ratio (OR) = .43, 95% CI 2-sided [.29 to .64]
Statistical Analysis 2: Comparison: Intervention: Teen Choices vs Comparison: Health In Motion; Test type: Superiority or Other; p = .003, Regression, Logistic; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = .47, 95% CI 2-sided [.29 to .77]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention: Teen Choices | Comparison: Health In Motion
Serious Adverse Events (participants affected / at risk) | 0/2000 | 0/1901
Other Adverse Events (participants affected / at risk) | 0/2000 | 0/1901

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes